CLINICAL TRIAL: NCT03036748
Title: Increased Activity of ENaC in Proteinuric Kidney Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Odense University Hospital (Other); Region of Southern Denmark (Other)
Responsible Party: Principal Investigator, Gitte Rye Hinrichs, Doctor, University of Southern Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ENaC activation
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Kidney Transplant; Complications
MeSH Terms: interventions — Diet; Amiloride

STUDY DESIGN:
Intervention Model Description: Experimental: Kidney transplant recipients with ACR > 300mg/g receiving standardized sodium diet (150 mmol NaCl/day) for 5 days and amiloride tablet 10 mg two times daily (morning and afternoon) on the last day.
  Interventions:◦Dietary Supplement: Standardized salt diet
  ◦Drug: Amiloride
  •Experimental: Kidney transplant recipient with ACR< 30mg/g (Control) receiving a standardized salt diet (150 mmol NaCl/day) for 5 days, then amiloride tablet 10 mg two times daily (morning and afternoon) for 1 day.
  Interventions:◦Dietary Supplement: Standardized salt diet
  ◦Drug: Amiloride
Masking Description: open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TX control (Experimental): Kidney transplant recipients with urinary albumin/creatinin-ratio < 30mg/g
  Interventions: Dietary Supplement: Standardized sodium diet; Drug: Tbl amiloride
- TX Proteinuria (Experimental): Kidney transplant recipients with urinary albumin/creatinin-ratio > 300mg/g
  Interventions: Dietary Supplement: Standardized sodium diet; Drug: Tbl amiloride

INTERVENTIONS:
Dietary Supplement: Standardized sodium diet — Dietary Supplement: Standardized salt diet 150 mmol NaCl per day given as three meals daily for 5 consecutive days.
  Other Names: Diet
Drug: Tbl amiloride — Drug: Amiloride Amiloride tablet 10 mg two times daily (morning and afternoon) for one day
  Other Names: Amiloride

SUMMARY:
The aim of this study is to determine if amiloride, a diuretic drug, is capable of increasing renal salt excretion, lowering blood pressure and inhibiting uPA in kidney transplant recipients with proteinuria compared to normoalbuminuric transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* One Group of kidney transplant recipients with ACR< 30mg/g
* One Group of kidney transplant recipients with ACR >300mg/g

Exclusion Criteria:

* Treatment with amiloride, spironolactone, aldosterone- or analogs or tranexamsyre
* Pregnancy
* Clinically relevant organic or systemic disease including malignancy
* eGFR or creatinin-clearance < 30ml/min
* hyperkalemia (s-potassium > 5,0mmol/l)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
24-hour urinary sodium excretion induced by amiloride | Change from baseline urinary sodium (after 4 days of standadized sodium diet) excretion at 24 hours after amiloride administration

SECONDARY OUTCOMES:
Office or 24h blood pressure measurements | Change from baseline office blood pressure at day 4 of salt diet and at 24 hours after amiloride administration

CONTACTS AND LOCATIONS:
Overall Officials: Gitte Rye Hinrichs, MD, PHD, Principal Investigator — Cardiovascular and Renal research
Locations (1):
- Odense University Hospital, Odense, Denmark

REFERENCES:
- [Derived] Isaksson GL, Hinrichs GR, Andersen H, Bach ML, Weyer K, Zachar R, Henriksen JE, Madsen K, Lund IK, Mollet G, Bistrup C, Birn H, Jensen BL, Palarasah Y. Amiloride Reduces Urokinase/Plasminogen-Driven Intratubular Complement Activation in Glomerular Proteinuria. J Am Soc Nephrol. 2024 Apr 1;35(4):410-425. doi: 10.1681/ASN.0000000000000312. Epub 2024 Jan 23. PMID 38254266